CLINICAL TRIAL: NCT04120259
Title: Effect of Apple Cider Vinegar and Metformin Combination vs Metformin Alone in Type 2 Diabetics:A Randomized Controlled Trial
Brief Title: Effect of Apple Cider Vinegar and Metformin Combination vs Metformin Alone in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr Momina Abid, Dr Momina Abid, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Acetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Intervention: Metformin Tablet oral 750 mg OD
  Interventions: Drug: Metformin Oral Tablet
- Group 2 (Experimental): Intervention: Metformin 750 mg oral plus 2 tablespoons of apple cider vinegar OD
  Interventions: Drug: Metformin Oral Tablet; Dietary Supplement: Vinegar

INTERVENTIONS:
Drug: Metformin Oral Tablet — A biguanide drug used as a first line therapy for Diabetes MellitusType 2
Dietary Supplement: Vinegar — A common herbal/dietary supplement used for centuries as an anti bacterial, cleaning,cooking, anti diabetic agent, to name a few uses.
  Arms: Group 2

SUMMARY:
'This study aims to compare the effect of Metformin alone vs Metformin plus Apple Cider Vinegar in newly diagnosed Type 2 Diabetic Patients

DETAILED DESCRIPTION:
Diabetes Mellitus is one of the oldest diseases known to men and has been treated with multiple agents,organic and with the current pharmacological advancement,with multiple synthetic drugs as well.

Metformin has been considered first line for the treatment of Type 2 Diabetes, however presents itself with a side effect profile of GI distress, Vitamin B12 deficiency,to name a few.

Vinegar has been used as therapeutic agent for centuries for multiple ailments including diabetes. This study aims to evaluate the combined effects of drug and natural therapy and compare it with conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed Type 2 diabetic patients taking metformin 750 mg daily as the oral antidiabetic agent
* Patients with Hemoglobin A1c in the range of 6.5 to 7.5%

Exclusion Criteria:

* All newly diagnosed Diabetic Patients requiring a dosage other than 750 mg per day
* Patients on Insulin Therapy or any drugs for diabetes other than Metformin
* Pregnant and Lactating women
* Patients with food allergies to either apple or any source of vinegar
* Patients unable to communicate efficiently\mentally challenged
* Type 2 Diabetic patients with any of the complications of long standing uncontrolled diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
BMI (Anthropometric Measurement) | 12 weeks
  Body Mass Index: A measure of obesity calculated as weight in kilograms divided by height in meters square
Measurement of Hemoglobin A1c | 12 weeks
  A blood test for Glycated Hemoglobin that represents a 2-3 month glycemic control
Measurement of Fasting Blood Sugar | 12 weeks
  A blood test that involves the measurement of plasma glucose after 8 to 12 hours of fasting

CONTACTS AND LOCATIONS:
Overall Officials: Dr Momina Abid, MBBS,M Phil (ongoing), Principal Investigator — Ziauddin University; Dr Zahida Memon, MBBS,M Phil,PhD, Principal Investigator — Ziauddin University
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No